CLINICAL TRIAL: NCT00005693
Title: Computer Assisted Instruction Weight Management for Low Literacy Populations
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4238; R01HL048064 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To develop and evaluate a computer assisted instruction (CAI) weight management program in an adult population with low literacy at Sheehan Memorial Hospital's Family Care Center (FCC), an outpatient clinic serving the inner city of Buffalo, New York.

DETAILED DESCRIPTION:
BACKGROUND:

This was the first study in patient care informatics in which nutrient analysis methodology was used on a day-to-day basis to motivate low literate individuals to improve their food choice behavior and physical activity. The deliverables of this investigation included revised and enhanced software, professional documentation, and a participant workbook. These materials were designed so that they could be integrated into any risk factor reduction program for low literacy populations.

DESIGN NARRATIVE:

The CAI featured voice recognition, giant cursor movement, and a graphics-based environment using pictures to facilitate an exceptionally easy to use and understand software program and booklet. The voice recognition technology was linked with compact disk read only memory (CD ROM) to visually display food choices and physical activities for ease of recording data by the individual. The software was formatted so that health professionals could select preference levels which corresponded to the motivational level of the individual. The four-session CAI intervention had two planned maintenance sessions. The output was personalized and in color. It was designed to identify problematic foods in the diet, improve food selections, and increase physical activity. Stars were printed for adherence to individual goals.

One hundred and fifty (150) men and 150 women, between age 20 and age 44, with a reading level of 8th grade or less, who were between 20 percent and 40 percent over their ideal body weight, were randomly assigned to three groups. The design compared a control group without the intervention, a group experiencing the CAI intervention and hands-on computer use, and a group experiencing the intervention but not the CAI component or computer use. All groups were pretested, posttested, and follow-up tested at six months and twelve months following baseline. The primary outcome measures were weight loss, nutrient intake, and physical activity. Data were analyzed using a two-way analysis of covariance and appropriate t-tests.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-04; Study Completion 1995-03 (Actual)